CLINICAL TRIAL: NCT06231719
Title: Evaluation of the Efficacy of Manual Pressure and Local Cold Spray Application in Reducing Pain Caused by Human Anti-D Immunoglobulin Injection in Pregnant Women: A Randomized Controlled Study
Brief Title: Efficacy of Manuel Pressure and Local Cold Spray in Reducing Injection Pain in Pregnant Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulsum Coskun (Other)
Responsible Party: Sponsor-Investigator, Gulsum Coskun, Principal Investigator Nurse, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Kartalsehir
Record Dates: First submitted 2023-11-30; First posted 2024-01-30 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Pain, Acute; Alloimmunisation in Pregnancy; Injection Site; Injection Fear
Keywords: Human Anti-D Immunglobulin; Red Blood Cell; Alloimmunization; Injection Pain; Local Cold Therapy; Manuel Pressure; Pregnancy
MeSH Terms: conditions — Acute Pain; Iatrophobia

STUDY DESIGN:
Intervention Model Description: Two intervention ,one control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anti-D Immunglobulin Injection with Cold Spray (Experimental): Using cold spray before the Anti-D immunoglobulin injection
  Interventions: Other: Cold Spray
- Anti-D Immunglobulin Injection with Manuel Pressure (Experimental): Apply Manuel pressure before the Anti-D immunoglobulin injection
  Interventions: Other: Manuel Pressure
- Standard Anti-D Immunoglobulin Injection (Placebo Comparator): Standard procedure for Anti-D immunglobulin injection
  Interventions: Other: Standard Injection Procedure

INTERVENTIONS:
Other: Cold Spray — Using cold spray for injection site before the Anti-D immunglobulin injection. 2 sprays of cold spray are applied from a distance of 25 cm.
  Arms: Anti-D Immunglobulin Injection with Cold Spray
Other: Manuel Pressure — Using manuel pressure ( about 10 second ) before the Anti-D immunglobulin injection.
  Arms: Anti-D Immunglobulin Injection with Manuel Pressure
Other: Standard Injection Procedure — Using any special method for injection
  Arms: Standard Anti-D Immunoglobulin Injection

SUMMARY:
A randomized controlled study was planned to determine the effect of manual pressure and local cold spray application on the intensity of pain, fear, hemodynamic parameters, and satisfaction related to the pain reduction of human Anti-D immunoglobulin injection administered to pregnant women.

DETAILED DESCRIPTION:
Injections are a commonly used treatment method that can induce fear, tension and anxiety in individuals despite their frequent use. The use of long needles, especially for intramuscular injections, to reach the target area through an injection can disrupt tissue integrity and cause discomfort. Therefore, injection pain is a widespread problem. Depending on the severity of perceived pain, it can affect an individual's hemodynamic parameters. Pain-related factors such as high heart rate, blood pressure, low oxygen saturation, and hyperventilation can develop. Primary caregivers, such as nurses, attempt to minimize pain by using pharmacological methods (local anesthesia, adjuvant analgesia, non-steroidal anti-inflammatory drugs (NSAID), opioids, paracetamol) and non-pharmacological interventions (manual pressure, cold application, Helfer skin tap, Shotblocker, massage, internal rotation, Buzzy). Human Anti-D immunoglobulin injection, like all other injections, causes pain, negatively affecting the quality of life and treatment experiences of individuals. In our study, we aim to evaluate the effectiveness of pre-injection manual pressure and local cold spray application, create data in the clinical field and reduce injection pain in pregnant women to have a positive impact on injection satisfaction and hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand, speak, read and understand Turkish
* Volunteering to participate in the study
* Being pregnant (gestational week 20 and above)
* Being between the ages of 18-45
* Has not had an IM injection in the last week
* There are no complications related to IM injections such as pain, abscess, infection, tissue necrosis, hematoma at the IM injection site.
* Not taking any analgesics before the procedure
* No chronic disease
* Those who do not have visual or cognitive impairments that prevent them from marking measurement tools

Exclusion Criteria:

* Not volunteering to participate in the study
* Having chronic pain disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Approximately 3 minute after injection
  Visual Analog Scale will be used to measure the injection pain intensity in pregnant women receiving the Human Immunoglobulin Anti-D injection. Participants in the study will be asked to mark their own pain level on a 10 cm ruler with "no pain" at one end and "unbearable pain" at the other. The preference for using VAS in pain intensity measurement is due to its ability to provide a numerical and replicable measurement according to the purpose.
Injection Satisfaction | Approximately 4 minute after injection
  When reviewing the literature, no specific scale for assessing satisfaction with IM injection applications was found. Upon examining national and international studies assessing satisfaction with IM injection, it was determined that VAS was utilized.In order to assess the satisfaction of patients after the injection, a scale with a vertical line of 10 cm, with "Very Satisfied" at one end and "Not Satisfied at All" at the other end, will be used. The selection of this scale is primarily influenced by its similarity to VAS and its ease of understanding and marking. The use of a vertical dimension is deemed appropriate for better clarity.
Pain Fear | Before injection
  The Pain Fear Scale III was developed by McNeil and Rainwater to measure fear and/or anxiety related to pain. Ünver and Turan conducted a Turkish validity and reliability study for the scale. The scale consists of three subscales, each with 10 items. The subscales and their respective items are listed. In evaluating the scale without reverse scoring, items are rated on a Likert-type scale ranging from 1 to 5 (1-Never, 2-Slightly, 3-Fairly, 4-Very, 5-Extremely). The minimum total score is 30, and the maximum total score is 150. For each subscale, the minimum score is 10, and the maximum score is 50. A higher score on the scale indicates higher pain fear.
Introductory Information Form | After participants agree to participate in the research and sign the informed consent form, this form is filled out by the researchers.All of these take approximately 15 minutes.
  The form prepared by the researcher, based on literature information, consists of a total of 10 questions related to the socio-demographic characteristics (age, height, weight, employment status, education level, job, blood type) and obstetric characteristics (last menstrual period, gravida , miscarriage, abortion, parity, type of delivery and previous use of Human Immunoglobulin Anti-D injection) of pregnant women prescribed with Human Immunoglobulin Anti-D injection. The same form will be used for recording the hemodynamic parameters (pulse rate, blood pressure, respiratory rate, and oxygen saturation) of pregnant women before and after the injection, which will be measured by the researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Coşkuner Potur, A. Professor, Study Director — Supervisor
Locations (1):
- Kartal Dr. Lütfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Detailed Information About Injection — https://www.rhogam.com/rhogam-science/

DOCUMENTS (1):
  • Informed Consent Form (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT06231719/ICF_000.pdf